CLINICAL TRIAL: NCT04528121
Title: Effect of CoDuSe Balance Training and Step Square Exercises on Risk of Fall in Multiple Sclerosis
Acronym: core stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lama Saad El-Din Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/002865
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: CoDuSe; balance; step square exercises; risk of fall; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: control group which received conventional selected exercise program in form of static and dynamic balance training exercises and study group received the same exercise training program in addition to CoDuSe balance training and step square exercises, three times per week for four weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): (CoDuSe) exercise inform of core stability, dual tasking, and sensory strategies the conventional selected exercise program inform of static and dynamic balance training exercises
  Interventions: Other: CoDuSe balance training and step square exercises; Other: conventional balance training
- control group (Experimental): the conventional selected exercise program inform of static and dynamic balance training exercises
  Interventions: Other: conventional balance training

INTERVENTIONS:
Other: CoDuSe balance training and step square exercises — The standardized intervention targeted visual, somatosensory, and vestibular aspects of balance and will be included with balance exercises
  Examples of core stability exercises as follows: in supine position with knees bent, slowly slide one heel forward to straighten leg; and, in four-point kneeling position, slide one foot in a straight line away from the body and lift the leg off the floor.
  Examples of dual-task exercises as walking while turning one's head and juggling a balloon.
  Examples of sensory strategies as standing and walking on uneven surfaces and standing with eyes closed.
  Arms: study group
Other: conventional balance training — static and dynamic balance training exercises from sitting, standing and ambulation activities

SUMMARY:
To investigate the effect of CoDuSe balance training and step square exercises on the risk of falls in multiple sclerosis. BACKGROUND: risk of fall & balance disabilities are considered serious problems in multiple sclerosis which results in loss of balance & physical inactivity.

………HYPOTHESES:

This study hypothesized that:

CoDuSe balance training and step square exercises will have a significant effect on the risk of falling in multiple sclerosis

RESEARCH QUESTION:

Is there an effect of CoDuSe balance training and step square exercises on risk of fall in multiple sclerosis?

DETAILED DESCRIPTION:
Fifty-two patients with multiple sclerosis will participate in this study.

The patients will randomly be divided into two equal groups; the control group which received the conventional selected exercise program and the study group received the same exercise training program in addition to CoDuSe balance training and step square exercises, three times per week for four weeks.

The Evaluation will done pre and post interventions included:

Biodex balance system (Risk falling), Short Physical Performance Battery (SPPB) & Morse Fall Scale.

ELIGIBILITY:
Inclusion Criteria:

* Fifty-two Remitting-relapsing multiple sclerosis RRMS patients,
* Age will range as (20:40) years old
* Illness duration not more than 10 years,
* with no relapses over the past three months,
* body mass index (25:35)

Exclusion Criteria:

* difficulty to communicate or to understand program instructions
* any other neurological deficits or orthopedic abnormalities,
* secondary musculoskeletal complication
* peripheral vestibulopathy, hepatic, renal, hemopoeitic, thyroid and cardiovascular diseases, cognitive dysfunction,
* hearing deficits, epilepsy or EEG abnormalities

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Biodex balance system | 4 weeks
  fast, accurate Fall Risk Screening and Conditioning Programme
Short Physical Performance Battery (SPPB) | 4 weeks
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests . It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people.
  The Short Physical Performance Battery (SPPB)test is designed to measure functional status and physical performance.
Morse Fall Scale | 4 weeks
  The Morse Fall Scale (MFS) is a rapid and simple method of assessing a patient's likelihood of falling A patient who scores under 25 points is considered to be at low risk of falling, a patient who scores between 25-45 points is considered to be at moderate risk of falling, and a patient who scores higher than 45 points is considered to be at high risk of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Lama S Mahmoud, Principal Investigator — Cairo University; Lama S Mahmoud, PHD, Principal Investigator — Lecturer,Department of physical therapy for Neuromuscular Disorders & its surgery / Faculty of physical therapy/ October 6 university; Hanan H Mohamed, PHD, Principal Investigator — Lecturer of physical therapy for neuromuscular disorders and its surgeries, modern university for technology & information (MTI) Egypt; Sobhy M Aly, PHD, Principal Investigator — Assistant professor, Department of Biomechanics, faculty of physical therapy, Cairo university
Locations (1):
- October 6 University, Giza, El-Sheikh Zayed City Giza 1133 Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No